CLINICAL TRIAL: NCT02529670
Title: Study of the Effect of Low Level Laser Therapy in the Dorsal Root Ganglion in the Diagnosis and Treatment of Chronic Low Back Pain
Brief Title: Low Level Laser Therapy in the Dorsal Root Ganglion in the Treatment of Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Vanessa Milanesi Holanda, MD, MS, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 53123716.3.0000.5511
Record Dates: First submitted 2015-08-11; First posted 2015-08-20 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Pain; Low Back Pain; Nociceptive Pain; Neuropathic Pain; Low Level Laser Therapy
Keywords: Low Level Laser Therapy; Low Back Pain; Diagnosis; Genetic; Clinical trial
MeSH Terms: conditions — Pain; Low Back Pain; Nociceptive Pain; Neuralgia; Disease | interventions — Lasers; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Laser (Experimental): 15 patients will be positioned in a prone horizontal position under anesthetic monitoring. The intervertebral foramen between the second and third lumbar vertebrae will be accessed by percutaneous puncture guided by fluoroscopy. Laser Photon III® (DCM) will be applied through fiber optics crossing G18 cannulas, during 84 seconds.
  Interventions: Procedure: Laser
- Radiofrequency (Active Comparator): 15 patients will receive radiofrequency in the second dorsal root ganglion through tubes G20, 150 mm long and 5 mm active tip in contact with the target, neuromodulation will be held for 300 seconds at 42oC.
  Interventions: Procedure: Radiofrequency
- Drug: Lidocaine (Active Comparator): In the local anesthetic group, 15 patients will receive the injection of 1 ml lidocaine without vasoconstrictor will be applied in the tubes G18, 150 mm long to block the second dorsal root ganglion.
  Interventions: Procedure: Drug: Lidocaine

INTERVENTIONS:
Procedure: Laser — Low level laser therapy will be delivered through Laser Photon III ® (DMC) in the second lumbar dorsal root ganglion.
  Arms: Laser
Procedure: Drug: Lidocaine — 1 mL of Lidocaine will be delivered in the second lumbar dorsal root ganglion through fluoroscopy.
  Arms: Drug: Lidocaine
Procedure: Radiofrequency — Radiofrequency will be delivered during 300 seconds, 42oC in the second lumbar dorsal root ganglion.
  Arms: Radiofrequency

SUMMARY:
Chronic axial low back pain is a public health problem and has a high socioeconomic impact. The dorsal ganglion of the second spinal nerve (GDL2) is a cluster of neuronal bodies responsible for sensory afferent inputs from more than 80% of the lumbar region. Low-level laser therapy (LLLT) is proven effective to help relieve pain. Thus, the aim of this project is to determine the effect of LLLT on GDL2 when applied to assist in the diagnosis and treatment of chronic axial low back pain. Methodology: 45 patients will be randomized into three groups: laser, radiofrequency and local anesthetic. The patient will be positioned in a prone horizontal position under anesthetic monitoring. The intervertebral foramen between the second and third lumbar vertebrae will be accessed by percutaneous puncture guided by fluoroscopy. In the local anesthetic group, injection of 1 ml lidocaine without vasoconstrictor will be applied in the tubes G20, 150 mm long and 5 mm active tip in contact with the target. In the radiofrequency group, neuromodulation will be held for 300 seconds at 42oC. In the laser group, the laser Photon III® (DCM) will be applied through optic fiber crossing G18 cannulas, during 84 seconds. The pain score will be assessed by visual analog scale. Temperature will be measured and aspirate periganglionic sample, trans-operatively, to study Interleucins-1β and TNF-alpha assessed by ELISA and genetic evaluation trough RNA seek, RNA isolation and ATP quantification. The data will be evaluated for normality and subjected to appropriate statistical analysis, in order to seek representation, as same as the level of significance of the studied samples.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain (more than 3 months of nociceptive or neuropathic pain).
* No neurological deficits

Exclusion Criteria:

* Active lumbar cancer
* Active infection
* Coagulation disorders

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Measure using Visual Analog Scale | 5 minutes before procedure
  Self reported pain intensity following Visual Analog Scale, scored 0-10 (0=no pain; 10=the worst pain ever).
Pain Intensity Measure using the change in Visual Analog Scale from baseline at 1 month | 5 minutes after procedure
  Patients will report the intensity of the pain using the score in visual analogue scale, scored 0-10 (0=no pain; 10=the worst pain ever).
Pain Intensity Measure using the Visual Analog Scale | 1 month and 6 months after procedure
  In follow up, patients will report the intensity of the pain using the score in visual analogue scale, scored 0-10 (0=no pain; 10=the worst pain ever).

SECONDARY OUTCOMES:
Immunochemistry to analyse IL-1, IL-10, TNF alfa. | Samples collected 1 minute after the application of laser, radiofrequency or lidocaine
  Through the needle used the sample will be collected and examined by immunocytochemical staining and ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- Nove de Julho Universtiy, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Rydevik BL, Myers RR, Powell HC. Pressure increase in the dorsal root ganglion following mechanical compression. Closed compartment syndrome in nerve roots. Spine (Phila Pa 1976). 1989 Jun;14(6):574-6. doi: 10.1097/00007632-198906000-00004. PMID 2749371
- [Background] Hart LG, Deyo RA, Cherkin DC. Physician office visits for low back pain. Frequency, clinical evaluation, and treatment patterns from a U.S. national survey. Spine (Phila Pa 1976). 1995 Jan 1;20(1):11-9. doi: 10.1097/00007632-199501000-00003. PMID 7709270
- [Background] Deyo RA, Mirza SK, Martin BI. Back pain prevalence and visit rates: estimates from U.S. national surveys, 2002. Spine (Phila Pa 1976). 2006 Nov 1;31(23):2724-7. doi: 10.1097/01.brs.0000244618.06877.cd. PMID 17077742
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934
- [Background] Frymoyer JW, Cats-Baril WL. An overview of the incidences and costs of low back pain. Orthop Clin North Am. 1991 Apr;22(2):263-71. PMID 1826550
- [Background] Katz JA. Getting the lowdown on back pain. Nursing. 2001 Dec;31(12):24. doi: 10.1097/00152193-200131120-00008. No abstract available. PMID 11921711
- [Background] Schaeffer V, Meyer L, Patte-Mensah C, Mensah-Nyagan AG. Progress in dorsal root ganglion neurosteroidogenic activity: basic evidence and pathophysiological correlation. Prog Neurobiol. 2010 Sep;92(1):33-41. doi: 10.1016/j.pneurobio.2010.04.009. Epub 2010 May 10. PMID 20438798
- [Background] de Souza Grava AL, Ferrari LF, Defino HL. Cytokine inhibition and time-related influence of inflammatory stimuli on the hyperalgesia induced by the nucleus pulposus. Eur Spine J. 2012 Mar;21(3):537-45. doi: 10.1007/s00586-011-2027-8. Epub 2011 Sep 25. PMID 21947908
- [Background] Chow R, Yan W, Armati P. Electrophysiological effects of single point transcutaneous 650 and 808 nm laser irradiation of rat sciatic nerve: a study of relevance for low-level laser therapy and laser acupuncture. Photomed Laser Surg. 2012 Sep;30(9):530-5. doi: 10.1089/pho.2012.3248. Epub 2012 Jul 10. PMID 22779441
- [Background] Lauria G, Bakkers M, Schmitz C, Lombardi R, Penza P, Devigili G, Smith AG, Hsieh ST, Mellgren SI, Umapathi T, Ziegler D, Faber CG, Merkies IS. Intraepidermal nerve fiber density at the distal leg: a worldwide normative reference study. J Peripher Nerv Syst. 2010 Sep;15(3):202-7. doi: 10.1111/j.1529-8027.2010.00271.x. PMID 21040142